CLINICAL TRIAL: NCT02399943
Title: Molecular Basket Trial In Multiple Malignancies With Common Target Pathway Aberrancies
Brief Title: A Trial of Trametinib and Panitumumab in RAS/RAF Wild Type Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOBILITY-001
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; KRAS Wildtype; NRAS Wildtype; BRAF Wildtype
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trametinib; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trametinib and Panitumumab (Experimental): Trametinib: 2 mg QD, orally, continuously.
  Panitumumab: 6 mg/kg, intravenously, Q2W
  Interventions: Drug: Trametinib; Drug: Panitumumab

INTERVENTIONS:
Drug: Trametinib
  Other Names: MEKINIST
Drug: Panitumumab
  Other Names: VECTIBIX

SUMMARY:
This is a phase 2 study (the second phase in testing a new drug or drug combination) to see how useful the combination of two drugs, panitumumab and trametinib, are in patients with advanced colorectal cancer with KRAS, NRAS, or BRAF wild type (genes that are not mutated).

Panitumumab is a drug that is approved by Health Canada for the treatment of advanced colorectal cancer with KRAS wild type. Panitumumab works by binding to and blocking the protein, epidermal growth factor receptor (EGFR) from working.

Trametinib is a drug that is approved by Health Canada for the treatment of melanoma with a mutation in the BRAF gene. Trametinib works by binding to and blocking mitogen-activated protein kinase kinase (MEK) 1 and MEK2 from working.

Previous studies have shown that the combination of panitumumab and trametinib may be more useful in KRAS, NRAS, or BRAF wild type colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* KRAS/NRAS/BRAF wild type colorectal cancer, not responsive to standard therapies, no approved or curative therapy, refuse standard therapy
* Prior 5-FU, oxaliplatin and irinotecan
* ECOG Performance Status of 0 or 1
* Able to swallow/retain oral drugs
* Able and agree to have provide tumor tissue/have biopsies
* Agree to use contraception
* Not pregnant
* Adequate organ system function

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapies <28 days or 5 half lives
* Prior EGFR, MEK, or RAF inhibitor or regorafenib
* Current use of prohibited medications
* Unresolved side effects
* GI disease or other condition affecting GI absorption
* Mucosal or internal bleeding
* Any major surgery <four weeks
* HIV, HBV, or HCV positive
* Active infection
* Leptomeningeal disease
* Brain metastases
* Unacceptable QTcF interval
* Significant uncontrolled arrhythmias
* Acute coronary syndromes, myocardial infarction, coronary angioplasty, or stenting or bypass grafting < 6 mos.
* Class II, III, or IV heart failure
* Other clinically significant ECGs
* Intra - cardiac defibrillators
* Cardiac metastases
* Condition that may interfere with patient safety
* Hypersensitivity to study drugs
* Severe or uncontrolled systemic diseases
* Pregnant or lactating
* Retinal vein occlusion
* Interstitial lung disease or pneumonitis
* Active liver or biliary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2019-04 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who experience complete response, partial response, or stable disease | 24 weeks
  by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Frequency and proportion of patients who experience side effects. | 3 years
  by system organ class and preferred term
Proportion of subjects achieving either a complete or partial tumor response | 3 years
  by RECIST 1.1 criteria
Time period from the first dose of Trametinib and Panitumumab to the first date in which progression or death is observed | 3 years
Date of first confirmed response to the first date in which progression is observed | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Alshammari K, Aung KL, Zhang T, Razak ARA, Serra S, Stockley T, Wang L, Nguyen J, Spreafico A, Hansen AR, Zwir D, Siu LL, Bedard PL. Phase II Trial of Trametinib and Panitumumab in RAS/RAF Wild Type Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2021 Dec;20(4):334-341. doi: 10.1016/j.clcc.2021.07.004. Epub 2021 Jul 24. PMID 34417144